CLINICAL TRIAL: NCT06690203
Title: TaichungVGH Taichung Veterans General Hospital
Brief Title: Evaluation of the Safety and Clinical Efficacy of NRICM102 in Patients With Chronic Lower Respiratory Tract Diseases
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Pin-Kuei Fu, MD, PhD, Director; Integrated Care Center of Interstitial Lung Disease (ICCILD), Taichung Veterans General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CF24327B
Record Dates: First submitted 2024-10-15; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Chronic Lower Respiratory Diseases
Keywords: Chronic lower respiratory diseases; NRICM102; Inflammation; safety; Biomarkers
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A. Combining NRICM102 decoction with standard treatment for 12 weeks (Other): Combining NRICM102 decoction with standard treatment for 12 weeks
  Interventions: Combination Product: NRICM102
- B. Combining NRICM102 decoction with standard treatment for 24 weeks (Other): Combining NRICM102 decoction with standard treatment for 24 weeks
  Interventions: Combination Product: NRICM102

INTERVENTIONS:
Combination Product: NRICM102 — A traditional Chinese medicine formula

SUMMARY:
This study is to assess safety and efficacy of NRICM102 decoction in participants with CLRD. This study will be conducted in 70 participants. The study consists of 3 periods: a 4-week screening period, a treatment period for at least 12 weeks up to 24 weeks.

DETAILED DESCRIPTION:
* Investigational product(s)： NRICM102 Decoction
* Development Phase: A real-world Prospective study
* Study Design：

  1. Experimental Group: Standard of care combined NRICM102 for 12weeks
  2. Blinding：Open
  3. Randomization: No
  4. Parallel design : Not applicable
  5. Treatment Period：12 to 24 weeks by groups
  6. Study Period: From 01/07/2024 to 31/12/2025
  7. Dose adjustment： Not applicable
  8. Study location： Single
* Study Procedures： This study is to assess safety and efficacy of NRICM102 decoction in participants with CLRD. This study will be conducted in 70 participants. The study consists of 3 periods: a 4-week screening period, a treatment period for at least 12 weeks up to 24 weeks. In principle, the two groups are divided into 1:1. The study group period is divided into a continuous treatment group and a discontinued treatment group. The purpose is to evaluate the drug safety of continuous treatment for 24 weeks and the similarities and differences in the physiological assessment of the subjects between the two groups, so as to serve as a reference for the design of a combined treatment program of traditional Chinese and Western medicine for chronic respiratory diseases. Since subjects may terminate early during the taking period, we also designed an evaluation time point, and also conducted an evaluation at the early end of time (EOS).
* Statistical Methods：

  1. Main study Hypothesis：Not applicable
  2. Estimated Sample Size：This study will be conducted in 70 participants. 50 subjects can be evaluated in the trial.
  3. Efficacy assessment group：Intent-to-treat (ITT)
  4. Interim analysis：No
  5. Statistical methods： All participants who have been randomized to study intervention and who have received at least one dose of study intervention will be included in the Efficacy Analysis Set. The Safety Analysis Set is defined as all participants who have been randomized to study intervention.

All results will be presented by treatment with descriptive statistics appropriate to the nature of the variables. Demographic and baseline characteristics will be presented as follows; for continuous variables, the number of non-missing observations, mean, standard deviation (SD), standard error (SE) of the mean, 95% confidence interval (CI) of the mean (except safety data), median, first and third quartiles, minimum and maximum, will be presented; for categorical variables: counts (n) and percentages (%) (where specified) will be presented. These summaries will be provided by time point of assessment as appropriate.

Details on the handling of missing data for the safety or efficacy analyses will be provided.

1. Safety will be assessed by descriptive analysis of vital signs, ECGs, laboratory assessments and AEs reported.
2. Change from baseline in health related QOL questionnaires ACT, ACQ-5, CAT, SGRQ and mMRC, spirometry and walking distance of visit and average over the treatment period will be reported, and subgroup analysis in CLRT will be provided at Weeks 4, 12, 24 and average over the treatment period.

   * 6. Handling of Missing Data： The missing data will not be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Diagnosed of chronic lower respiratory tract disorder(such as : asthma, COPD, emphysema, chronic bronchitis, bronchiectasis, lung fibrosis) by pulmonologist
* Have symptom of chronic cough, cough with sputum after using of a maintenance respiratory medication and stable disease more than 3 months.
* Willing to be evaluated by a Traditional Chinese Physician whether use of NRICM102 is suitable.
* The patient can use NRICM102 therapy after Traditional Chinese Physician evaluate. Able to understand and sign an informed consent ( or have a legal representative who is able to do so)

Exclusion Criteria:

* Females who are breastfeeding or pregnant at screening.
* Life threatening (e.g. intensive care admission and/or use of mechanical ventilation) respiratory failure event in the past 3 months.
* Patients with gastrointestinal malabsorption or condition that might affect the absorption of NRICM102 in the opinion of investigator. (exp: Irritable bowel syndrome, acute gastritis, duodenal ulcer..).
* Acute exacerbation or unstable vital signs on screening stage.
* Patient who have malignancy and receiving chemotherapy/ target therapy at screening.
* Diagnosis of liver cirrhosis or active hepatitis infection.
* Patient having renal dysfunction with Creatinine Clearance Calculator (CCR) < 30mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of combining NRICM102 decoction with standard treatment for 12 to 24 weeks in subjects comorbid with chronic respiratory diseases to treat the chronic respiratory symptoms | Up to study completion approximately 24 weeks
  The proportion of AE and/or SAE with grading.

SECONDARY OUTCOMES:
Asthma control test (ACT) for asthma patients among different treatment periods (12 or 24 weeks) | Up to study completion approximately 24 weeks
Asthma Control Questionnaire (ACQ)-5 for asthma patients among different treatment periods (12 or 24 weeks) | Up to study completion approximately 24 weeks
The COPD Assessment Test (CAT) among different treatment periods (12 or 24 weeks) | Up to study completion approximately 24 weeks
St. George's Respiratory Questionnaire (SGRQ) among different treatment periods (12 or 24 weeks) | Up to study completion approximately 24 weeks
  St. George's Respiratory Questionnaire (SGRQ)
modified Medical Research Council (mMRC) scale among different treatment periods (12 or 24 weeks) | Up to study completion approximately 24 weeks
  modified Medical Research Council (mMRC) scale
Body Constitution Questionnaire (BCQ) in traditional Chinese medicine among different treatment periods (12 or 24 weeks) | Up to study completion approximately 24 weeks
  Body Constitution Questionnaire (BCQ) in traditional Chinese medicine

CONTACTS AND LOCATIONS:
Overall Officials: Pin-Kuei Fu, Principal Investigator — chairman; Integrated Care Center of Interstitial Lung Disease (ICCILD)
Locations (1):
- Taichung Veterans General Hospita, Taichung, No.1650, Taiwan Boulevard Sect. 4, Taiwan

IPD SHARING:
Plan to Share IPD: No